CLINICAL TRIAL: NCT00911820
Title: A Randomized, Multicenter, Phase II Trial of Cisplatin, Irinotecan and Bevacizumab (PCA) vs. Docetaxel, Cisplatin, Irinotecan and Bevacizumab (TPCA) in Metastatic Esophageal and Gastric Cancer
Brief Title: Cisplatin, Irinotecan and Bevacizumab (PCA) Versus Docetaxel, Cisplatin, Irinotecan and Bevacizumab (TPCA) in Metastatic Esophageal and Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); SCRI Development Innovations, LLC (Other); Texas Oncology Cancer Center (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Peter C. Enzinger, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-039
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Esophageal Cancer; Gastric Cancer; Stomach Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Bevacizumab; Cisplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: PCA (Active Comparator): Patients first received bevacizumab 10 mg/kg IV on day 1 of every cycle (cycle length=21 days) at approximately 0.5 mg/kg/minute. Additionally, on days 1 and 8 of each cycle, patients received cisplatin 30 mg/m2 IV over 30 minutes and then irinotecan 65 mg/m2 IV over 30 minutes of each 3-week cycle. Treatment could continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Bevacizumab; Drug: Cisplatin; Drug: Irinotecan
- Arm B: TPCA (Active Comparator): Patients first received bevacizumab 10 mg/kg IV on day 1 of every cycle (cycle length=21 days) at approximately 0.5 mg/kg/minute. Additionally on days 1 and 8 of each cycle, patients received docetaxel 30 mg/m2 IV over 30 minutes followed by cisplatin 25 mg/m2 IV over 30 minutes and then irinotecan 50 mg/m2 IV over 30 minutes of each 3-week cycle.
  Interventions: Drug: Cisplatin; Drug: Irinotecan; Device: Docetaxel

INTERVENTIONS:
Drug: Bevacizumab
  Other Names: Avastin
  Arms: Arm A: PCA
Drug: Cisplatin
  Other Names: Platinol-AQ; Platinol
Drug: Irinotecan
  Other Names: Camptosar
Device: Docetaxel
  Other Names: Taxotere; Docefrez
  Arms: Arm B: TPCA

SUMMARY:
There is no clear standard of care for metastatic stomach or esophageal cancer in the United States. The purpose of this research study is to determine the differences between two regimens of chemotherapy; Arm A: PCA (Cisplatin, Irinotecan and Bevacizumab) and Arm B: TPCA (Docetaxel, Cisplatin, Irinotecan and Bevacizumab). Docetaxel, Cisplatin, and Irinotecan are traditional chemotherapy drugs. Bevacizumab is an antibody (a protein that attacks a foreign substance in the body). Bevacizumab is believed to stop the formation of new blood vessels that carry nutrients to tumors. Both of the chemotherapy regimens (PCA and TPCA) have been studied in patients with esophageal and gastric cancer, and we are trying to determine if one regimen will keep your cancer from growing and improve how long you can live.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate progression-free survival at 7 months in metastatic esophageal and gastric patients treated with either PCA or TPCA

Secondary

* To determine overall survival
* To determine the response rate (RECIST) in measurable disease patients
* To evaluate type and severity of toxicities associated with each regimen

Exploratory:

* To correlate expression of tumoral and serum VEGF with response and survival
* To correlate TGF alpha levels and tumor microvessel density with clinical activity of the combination of PCA or TPCA
* To examine circulating endothelial cells (CECs) as surrogate markers of antitumor activity of bevacizumab
* To explore if 7/7 and 7/6 UGT1A1 polymorphisms correlate with grade III/IV irinotecan-related diarrhea and neutropenia when irinotecan is given at relatively low dose to patients with esophageal and gastric cancer

DESIGN:

This trial was designed to compare 7-month progression-free survival between arms. The hypothesis was that TPCA would have superior outcome over PCA (70% vs 50%). With 40 eligible patients per arm followed for 1 year there was 80% power to detect a hazard ratio of 0.48 using the log-rank test at a one-sided type I error rate of 5%. Stratification factors were ECOG performance status 0/1 vs 2 and site of primary tumor (gastric vs GE junction/esophageal).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, unresectable esophageal, GE junction or gastric adenocarcinoma (including adenosquamous, or undifferentiated carcinoma). Measurable disease is not required.
* 18 years of age or older
* ECOG Performance Status=2
* Life expectancy of 12 weeks or greater
* Adequate bone marrow, renal and liver function as outlined in the protocol.
* Men and women of childbearing potential must use adequate contraception

Exclusion Criteria:

* Prior chemotherapy (except as part of pre- or post-operative therapy, completed at least 1 prior to start of this protocol).
* Squamous cell carcinoma histology of esophageal, GE junction or gastric tumor
* Known history of allergy or hypersensitivity to Chinese hamster ovary products, polysorbate 80, or any of the study drugs
* Treatment or planned participation in an experimental drug study within 4 weeks of C1 D1. Concurrent use of herbal medications or other alternative therapies
* Major surgical procedures, such as fine needle aspirations, port-a-cath placement, or core biopsies, within 7 days of cycle 1 day 1
* Palliative radiation to 25% or less of bone marrow, must be completed > 2 weeks prior to day 1, palliative radiation to > 25% of bone marrow, must be completed > 4 weeks prior to day 1
* Myocardial infarction, unstable angina, CVA or TIA or other thrombotic event in the past six months
* Inadequately controlled hypertension (defined as systolic blood pressure of >150mmHg and/or diastolic blood pressure of > 100mmHg). Initiation of antihypertensive medication is recommended, however adequate control of blood pressure must be documented prior to C1 D1
* No history of prior hypertensive crisis or hypertensive encephalopathy
* NYHA Grade II or greater congestive heart failure
* Clinically significant peripheral vascular disease
* Active bleeding from primary tumor
* Evidence of bleeding diatheses or coagulopathy (other than deep venous thrombosis, portal vein thrombosis, pulmonary embolism, or atrial fibrillation). Patients on therapeutic anticoagulation may be enrolled provided they have been clinically stable on anticoagulation for a least 2 weeks prior to C1 D1.
* Uncontrolled serious medical or psychiatric illness
* Uncontrolled diarrhea
* Peripheral neuropathy
* No known brain or other CNS metastasis by history or clinical examination
* Other active malignancy other than non-melanoma skin cancer or in-situ cervical carcinoma. A resected or previously treated cancer (other than in-situ carcinoma) must have demonstrated no evidence of recurrence for at least 3 years
* Urine protein:creatinine ratio 1.0 or greater at screening
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess with 6 months of C1 D1
* Serious, non-healing wound, ulcer or bone fracture
* Pregnant or breast feeding
* Inability to comply with study and/or follow-up procedures
* History of HIV seropositivity, hepatitis C virus, acute or chronic hepatitis B, or other serious chronic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter C. Enzinger, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology Research, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between July 2009 and April 2011.
Period: Overall Study
Arm/Group | Arm A: PCA | Arm B: TPCA
Started | 45 | 43
Treated | 44 (Randomized patients not treated: unable to confirm pathology (n=1)) | 41 (Randomized patients not treated: withdrew consent (n=2))
Completed (Since treatment was not of fixed duration, all patients were considered as 'Not Completed'.) | 0 | 0
Not Completed | 45 | 43
Not completed — RECIST progression | 12 | 8
Not completed — Adverse Event | 8 | 8
Not completed — Clinical Progression | 7 | 5
Not completed — Physician Decision | 5 | 9
Not completed — Decline in Performance Status | 4 | 2
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Death | 1 | 2
Not completed — Pursue surgery | 1 | 1
Not completed — Pursue Radiation | 1 | 0
Not completed — Still on Therapy | 2 | 2
Not completed — Pathology Not Confirmed | 1 | 0
Not completed — Withdraw before Receive Treatment | 0 | 2

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all treated patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: PCA | Arm B: TPCA | Total
Number analyzed (Participants) | 44 | 41 | 85
Age, Continuous [Median (Full Range); unit: years] | 59 [41 to 79] | 61 [40 to 85] | 60 [40 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 36 | 34 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 41 | 39 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44 | 41 | 85
ECOG Performance Status (PS) [Count of Participants; unit: Participants] — ECOG PS0: Fully active, able to carry on all pre-disease performance without restriction ECOG PS1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature ECOG PS2: Ambulatory and capable of all self-care but unable to carry out any work activities; Up and about more than 50% of waking hours
  Participants
    ECOG PS 0/1 | 43 | 40 | 83
    ECOG PS 2 | 1 | 1 | 2
Tumor Location [Count of Participants; unit: Participants]
  Esophagus | 20 | 17 | 37
  GE Junction | 9 | 12 | 21
  Gastric | 15 | 12 | 27

OUTCOME MEASURES:

1. Primary Outcome: 7-month Progression-Free Survival
Description: 7-month progression-free survival is the probability of patients remaining alive and progression-free at 7-months from study entry estimated using Kaplan-Meier methods. Per RECIST 1.0 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 2 cycles on treatment; Relevant for this endpoint was disease status at 7 months of follow-up.
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Arm A: PCA | Arm B: TPCA
Number analyzed (Participants) | 44 | 41
probability | 0.581 [0.421 to 0.712] | 0.582 [0.410 to 0.719]

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from study entry to death or date last known alive and estimate using Kaplan-Meier (KM) methods.
Time Frame: Patients in the study cohort were followed up to approximately 2.5 years as of this analysis.
Population: The analysis dataset is comprised of all treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: PCA | Arm B: TPCA
Number analyzed (Participants) | 44 | 41
months | 11.7 [9.6 to 15.4] | 13.4 [11.5 to 16.1]
Statistical Analysis 1: Comparison: Arm A: PCA vs Arm B: TPCA; Test type: Superiority; p = 0.714, Log Rank

3. Secondary Outcome: Best Response
Description: Best response on treatment was based on RECIST 1.0 criteria: Complete Response (CR) is complete disappearance of all target lesions; Partial Response (PR) is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. Both require confirmation no fewer than 4 weeks apart. CR/PR assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions. Progressive disease (PD) is at least a 20% increase in the sum of longest diameter of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions. Stable disease is defined as any condition not meeting above criteria.
Time Frame: Disease was evaluated radiologically at baseline and every 2 cycles on treatment; Treatment duration was a median of 5 cycles (up to approximately 1 year) in this study cohort as of this analysis..
Population: The analysis dataset is comprised of all treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: PCA | Arm B: TPCA
Number analyzed (Participants) | 44 | 41
Participants
  Complete Response | 3 | 0
  Partial Response | 22 | 21
  Stable Disease | 15 | 14
  Progressive Disease | 1 | 0
  Removed Before Restaging | 3 | 6

4. Secondary Outcome: Overall Response (OR) Rate
Description: Overall response (OR) rate was defined as achieving partial response (PR) or complete response (CR) based on RECIST 1.0 criteria on treatment. Per RECIST 1.0 for target lesions, CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. To be assigned a status of CR or PR, changes in tumor measurements must be confirmed by repeat assessments performed no fewer than 4 weeks after the response criteria are first met. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: as for outcome 3
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Arm A: PCA | Arm B: TPCA
Number analyzed (Participants) | 44 | 41
proportion of patients | .568 [.41 to .717] | .512 [.351 to .671]
Statistical Analysis 1: Comparison: Arm A: PCA vs Arm B: TPCA; Test type: Superiority; p = 0.605, Fisher Exact

5. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) requiring removal from the study or death. Patients alive and progression-free at last follow-up are censored. Per RECIST 1.0 criteria: progressive disease is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 2 cycles on treatment; Patients were followed for up to 2.5 years as of this analysis.
Population: The analysis dataset is comprised of all treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: PCA | Arm B: TPCA
Number analyzed (Participants) | 44 | 41
months | 7.9 [6.1 to 10.1] | 8.4 [6.2 to 9.7]
Statistical Analysis 1: Comparison: Arm A: PCA vs Arm B: TPCA; Test type: Superiority; p = 0.721, Log Rank

ADVERSE EVENTS:
Time Frame: Adverse events were assessed weeks 1 and 2 each cycle throughout treatment.Treatment duration was a median of 5 cycles (up to approximately 2 years) in this study cohort as of this analysis.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. All remaining events regardless of treatment attribution were classified as Other AEs. No further data is available to specify classification of other beyond the general term.
Arm/Group | Arm A: PCA | Arm B: TPCA
All-Cause Mortality (participants affected / at risk) | 0/44 | 3/41
Serious Adverse Events (participants affected / at risk) | 32/44 | 36/41
Other Adverse Events (participants affected / at risk) | 44/44 | 39/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: PCA (N=44) | Arm B: TPCA (N=41)
Abdomen, pain (Gastrointestinal disorders) | 0 | 2
Allergic reaction (Immune system disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 4
Back, pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cardiac troponin I (cTnI) (Investigations) | 1 | 0
Cardiac-ischemia (Cardiac disorders) | 1 | 0
CNS cerebrovascular ischemia (Nervous system disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Death - sudden death (General disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 6 | 5
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 10 | 13
Dizziness (Nervous system disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Esophagus, hemorrhage (Gastrointestinal disorders) | 0 | 1
Extremity-lower (gait/walking) (General disorders) | 1 | 0
Fatigue (General disorders) | 7 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3
GI-other (Gastrointestinal disorders) | 1 | 1
Head/headache (Nervous system disorders) | 1 | 1
Hematologic-other (Blood and lymphatic system disorders) | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 5 | 3
Hemorrhage-other (Vascular disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 3
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 1
Ileum, hemorrhage (Gastrointestinal disorders) | 0 | 1
Infection Gr0-2 neut, esophagus (Infections and infestations) | 1 | 0
Infection Gr0-2 neut, sinus (Infections and infestations) | 0 | 1
Infection w/ gr 3-4 neut, blood (Infections and infestations) | 1 | 0
Infection w/ gr3-4 neut, lung (Infections and infestations) | 1 | 0
Infection w/ gr3-4 neut, upper airway (Infections and infestations) | 0 | 1
Infection w/ gr3-4 neut, wound (Infections and infestations) | 1 | 0
Infection w/ unk ANC appendix (Infections and infestations) | 0 | 1
Infection-other (Infections and infestations) | 1 | 0
Leak, incl. anastomotic, small bowel (Injury, poisoning and procedural complications) | 0 | 1
Leukocytes (Investigations) | 6 | 11
Lymphopenia (Investigations) | 4 | 6
Nausea (Gastrointestinal disorders) | 4 | 5
Neutrophils (Investigations) | 11 | 13
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Perforation, colon (Gastrointestinal disorders) | 0 | 2
Platelets (Investigations) | 2 | 2
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 3
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Upper GI, hemorrhage NOS (Gastrointestinal disorders) | 2 | 0
Vascular access,Thrombosis/embolism (Injury, poisoning and procedural complications) | 1 | 1
Vomiting (Gastrointestinal disorders) | 4 | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: PCA (N=44) | Arm B: TPCA (N=41)
Abdomen, pain (Gastrointestinal disorders) | 17 | 19
Agitation (Psychiatric disorders) | 2 | 1
Alkaline phosphatase (Investigations) | 5 | 5
Allergic reaction (Immune system disorders) | 1 | 5
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Allergy-other (Immune system disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 17
ALT, SGPT (Investigations) | 1 | 6
Anorexia (Metabolism and nutrition disorders) | 19 | 28
Anus, hemorrhage (Gastrointestinal disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 9 | 10
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
AST, SGOT (Investigations) | 3 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 2
Back, pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Bicarbonate (Metabolism and nutrition disorders) | 1 | 1
Bilirubin (Investigations) | 1 | 3
Bone, pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 1
Buttock, pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cardiac-other (Cardiac disorders) | 2 | 2
Cataract (Eye disorders) | 1 | 0
Chelitis (Gastrointestinal disorders) | 1 | 0
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Chest/thoracic pain NOS (General disorders) | 5 | 3
Coagulation-other (Investigations) | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 1
Colon, hemorrhage (Gastrointestinal disorders) | 0 | 1
Confusion (Psychiatric disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 21 | 18
Constitutional, other (General disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Creatinine (Investigations) | 12 | 5
Cystitis (Renal and urinary disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 15 | 14
Depression (Psychiatric disorders) | 6 | 6
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 31 | 29
Distention/bloating, abdominal (Gastrointestinal disorders) | 0 | 2
Dizziness (Nervous system disorders) | 12 | 10
Double vision (Eye disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 7
Dyspepsia (Gastrointestinal disorders) | 7 | 6
Dysphagia (Gastrointestinal disorders) | 11 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Edema head and neck (General disorders) | 0 | 1
Edema limb (General disorders) | 5 | 3
Endocrine-other (Endocrine disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 2
Esophagitis (Gastrointestinal disorders) | 2 | 1
Esophagus, hemorrhage (Gastrointestinal disorders) | 1 | 0
Esophagus, pain (Gastrointestinal disorders) | 3 | 2
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Extremity-lower (gait/walking) (General disorders) | 1 | 0
Fatigue (General disorders) | 35 | 34
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Fever w/o neutropenia (General disorders) | 3 | 5
Flatulence (Gastrointestinal disorders) | 5 | 3
Flushing (Vascular disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 2 | 1
GI-other (Gastrointestinal disorders) | 6 | 9
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Head/headache (Nervous system disorders) | 18 | 12
Hearing-other (Ear and labyrinth disorders) | 1 | 0
Hematologic-other (Blood and lymphatic system disorders) | 1 | 0
Hematoma (Vascular disorders) | 2 | 1
Hemoglobin (Blood and lymphatic system disorders) | 34 | 28
Hemorrhage-other (Vascular disorders) | 1 | 1
Hemorrhoids (Gastrointestinal disorders) | 1 | 1
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Hot flashes (Vascular disorders) | 1 | 2
Hypercholesterolemia (Investigations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 20 | 18
Hyperkalemia (Metabolism and nutrition disorders) | 10 | 11
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 14 | 7
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 | 13
Hypocalcemia (Metabolism and nutrition disorders) | 9 | 15
Hypoglycemia (Metabolism and nutrition disorders) | 5 | 3
Hypokalemia (Metabolism and nutrition disorders) | 10 | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 13 | 16
Hyponatremia (Metabolism and nutrition disorders) | 15 | 14
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 5
Hypotension (Vascular disorders) | 5 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Infection Gr0-2 neut, anal/perianl (Infections and infestations) | 0 | 1
Infection Gr0-2 neut, catheter (Infections and infestations) | 1 | 1
Infection Gr0-2 neut, dental-tooth (Infections and infestations) | 1 | 2
Infection Gr0-2 neut, esophagus (Infections and infestations) | 0 | 1
Infection Gr0-2 neut, external ear (Infections and infestations) | 0 | 1
Infection Gr0-2 neut, foreign body (Infections and infestations) | 1 | 1
Infection Gr0-2 neut, oral cavity (Infections and infestations) | 0 | 0
Infection Gr0-2 neut, sinus (Infections and infestations) | 2 | 0
Infection Gr0-2 neut, skin (Infections and infestations) | 0 | 2
Infection Gr0-2 neut, ungual (Infections and infestations) | 0 | 1
Infection Gr0-2 neut, upper airway (Infections and infestations) | 1 | 2
Infection Gr0-2 neut, vagina (Infections and infestations) | 1 | 0
Infection w/ gr3-4 neut, paranasal (Infections and infestations) | 0 | 1
Infection w/ unk ANC colon (Infections and infestations) | 0 | 1
Infection w/ unk ANC lung (Infections and infestations) | 1 | 0
Infection w/ unk ANC prostate (Infections and infestations) | 0 | 1
Infection w/ unk ANC sinus (Infections and infestations) | 1 | 0
Infection w/ unk ANC skin (cellulitis) (Infections and infestations) | 1 | 0
Infection w/ unk ANC stomach (Infections and infestations) | 1 | 0
Infection w/ unk ANC upper airway NOS (Infections and infestations) | 1 | 0
Infection w/ unk ANC urinary tract NOS (Infections and infestations) | 1 | 0
Infection w/ unk ANC vagina (Infections and infestations) | 1 | 0
Infection-other (Infections and infestations) | 2 | 2
Injection site reaction (General disorders) | 0 | 1
INR (Investigations) | 0 | 1
Insomnia (Psychiatric disorders) | 8 | 10
Irregular menses (Reproductive system and breast disorders) | 0 | 1
Joint, pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Kidney, hemorrhage (Renal and urinary disorders) | 0 | 1
Leak, incl. anastomotic, esophagitis (Injury, poisoning and procedural complications) | 1 | 0
Leak, incl. anastomotic, small bowel (Injury, poisoning and procedural complications) | 0 | 2
Leukocytes (Investigations) | 23 | 23
Libido (Psychiatric disorders) | 0 | 1
Lip, pain (Gastrointestinal disorders) | 1 | 0
Lung, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lymphopenia (Investigations) | 6 | 6
Memory impairment (Nervous system disorders) | 1 | 1
Mental status (Nervous system disorders) | 1 | 1
Metabolic/Laboratory-other (Investigations) | 0 | 1
Middle ear, pain (Ear and labyrinth disorders) | 0 | 2
Muco/stomatitis (symptom) larynx (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 1 | 5
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 1 | 5
Muscle, pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscular/skeletal hypoplasia (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 3 | 4
Nail changes (Skin and subcutaneous tissue disorders) | 1 | 4
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 35 | 31
Neck, pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Neurologic-other (Nervous system disorders) | 1 | 2
Neuropathy CN I smell (Nervous system disorders) | 0 | 1
Neuropathy CN V jaw / face-sensory (Nervous system disorders) | 0 | 1
Neuropathy CN VII face-motor / taste (Nervous system disorders) | 0 | 1
Neuropathy-motor (Nervous system disorders) | 0 | 1
Neuropathy-sensory (Nervous system disorders) | 8 | 13
Neutrophils (Investigations) | 19 | 17
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 0 | 2
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 2 | 9
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 16 | 17
Obstruction, small bowel NOS (Gastrointestinal disorders) | 1 | 0
Ocular-other (Eye disorders) | 1 | 1
Oral cavity, hemorrhage (Gastrointestinal disorders) | 1 | 0
Oral cavity, pain (Gastrointestinal disorders) | 0 | 3
Oral gums, pain (Gastrointestinal disorders) | 0 | 2
Pain-other (General disorders) | 4 | 6
Palpitations (Cardiac disorders) | 1 | 1
Pelvic, pain (Reproductive system and breast disorders) | 1 | 1
Perforation, colon (Gastrointestinal disorders) | 0 | 2
Perforation, stomach (Gastrointestinal disorders) | 0 | 1
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Platelets (Investigations) | 23 | 17
Pleura, pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 2
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 | 2
PTT (Investigations) | 0 | 2
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 6
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 | 1
Rectum, hemorrhage (Gastrointestinal disorders) | 4 | 2
Rectum, pain (Gastrointestinal disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Renal/GU-other (Renal and urinary disorders) | 0 | 2
Rigors/chills (General disorders) | 4 | 2
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Skin-other (Skin and subcutaneous tissue disorders) | 3 | 1
Speech impairment (Nervous system disorders) | 1 | 0
Stenosis (incl anastomotic) esophagus (Gastrointestinal disorders) | 0 | 1
Stomach, pain (Gastrointestinal disorders) | 8 | 3
Sweating (Skin and subcutaneous tissue disorders) | 3 | 3
Syncope (Nervous system disorders) | 0 | 1
Taste disturbance (Nervous system disorders) | 8 | 15
Tearing (Eye disorders) | 0 | 3
Teeth (Gastrointestinal disorders) | 0 | 1
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0
Tremor (Nervous system disorders) | 1 | 6
Ulcer, cecum (Gastrointestinal disorders) | 0 | 1
Ulcer, colon (Gastrointestinal disorders) | 0 | 1
Ulcer, esophagus (Gastrointestinal disorders) | 0 | 1
Ulcer, gastric (Gastrointestinal disorders) | 0 | 1
Ulcer, stoma (Injury, poisoning and procedural complications) | 0 | 1
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Urinary frequency/urgency (Renal and urinary disorders) | 1 | 4
Urinary retention (Renal and urinary disorders) | 2 | 0
Vaginal mucositis (Reproductive system and breast disorders) | 1 | 0
Vascular access,Thrombosis/embolism (Injury, poisoning and procedural complications) | 0 | 1
Vascular-Other (Vascular disorders) | 0 | 1
Vision-blurred (Eye disorders) | 5 | 1
Vision-flashing lights/floaters (Eye disorders) | 1 | 0
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Vomiting (Gastrointestinal disorders) | 22 | 21
Weight gain (Investigations) | 1 | 0
Weight loss (Investigations) | 15 | 13
Wound - non-infectious (Injury, poisoning and procedural complications) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No